CLINICAL TRIAL: NCT00370461
Title: Basic Life Support Termination of Resuscitation in the Prehospital Environment for Primary Care Paramedics - A Prospective Observational Study of the Implementation of a Clinical Prediction Rule
Brief Title: Basic Life Support Termination of Resuscitation Implementation Study
Status: Completed | Type: Observational
Sponsor: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Laurie Morrison, Clinician Scientist, Sunnybrook Health Sciences Centre
Other Study IDs: MOP67110
Record Dates: First submitted 2006-08-29; First posted 2006-08-31 (Estimated); Last update posted 2015-11-17 (Estimated); Status verified 2015-11

CONDITIONS: Cardiac Arrest
Keywords: Basic Cardiac Life Support; Termination of Resuscitation; Emergency Medical Services; Primary Care Paramedics; Out of Hospital Cardiac Arrest
MeSH Terms: conditions — Heart Arrest; Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In Ontario, most people who experience a cardiac arrest at home (when their heart stops beating) only receive basic life support from Primary Care Paramedics (PCPs) and all are transported to the hospital. Most are pronounced dead by the emergency physician as the mean survival rate for these patients is 5%. Allowing Primary Care Paramedics to use a termination of resuscitation guideline would identify futile cases for which further resuscitation is unwarranted and decrease the number of patients being transported to the emergency department (ED) for pronouncement.

There are numerous advantages to this strategy; first, it may improve the efficiency of the ED because cardiac arrest patients require immediate attention that is diverted from patients who have a better chance at survival. Second, the risk of injury and the monetary costs for the paramedic and the public would be minimized with fewer "light and sirens" transports which are known to be hazardous to motorists, pedestrians, and Emergency Medical Services (EMS) personnel.

For each cardiac arrest, PCPs will respond to the call as usual and implement standard basic life support cardiac arrest protocols. Patients are then categorized according to the termination of resuscitation recommendations:

1. no return of spontaneous circulation is achieved (no heartbeat);
2. no shock was given prior to transport; and
3. the arrest (when the heart stops beating) was not witnessed by EMS personnel.

If all of these criteria are true, the PCP will contact the hospital and the decision by the emergency physician will then be made to stop life saving measures (terminate resuscitation) in the home or continue with life support and transport the patient to the local emergency department.

This study aims to document the usefulness of the termination of the resuscitation guideline in decreasing the rate of transport of out-of-hospital cardiac arrest patients to the ED. Secondary aims of this implementation study will be to describe the rates of erroneous application of the guideline. The comfort of use of the rule among paramedics and base hospital emergency physicians will be described.

DETAILED DESCRIPTION:
In Ontario, most victims of out-of-hospital cardiac arrest (OHCA) do not receive Advanced Cardiac Life Support (ACLS); rather, they receive only Basic Life Support (BLS) from Primary Care Paramedics (PCPs), where the survival rate is approximately 5%. Every one of these patients is transported to the Emergency Department (ED), where the vast majority are pronounced dead. Conversely, patients who do not respond to ACLS by Advanced Care Paramedics (ACPs) are pronounced dead in the field via patching to the Base Hospital Physician (BHP). Implementation of a termination of resuscitation (TOR) guideline for the PCP's use would decrease the number of non-viable patients transported to the ED.

A reduction of unsuccessfully resuscitated cardiac arrest patients transported to the ED would have numerous advantages. First, it may improve the efficiency of the ED health care system because cardiac arrest patients in the ED require immediate attention that is diverted from potentially more salvageable patients. Second, the risk of injury and the monetary costs for the paramedic and the public would be minimized with fewer "light and sirens" transports which are known to be hazardous to motorists, pedestrians, and EMS personnel. Additionally, it is less expensive to pronounce non-viable patients in the field. And, finally termination of resuscitative efforts in the field permits the paramedic to turn his attention and skill set to supporting the family through the initial stages of grief.

The most recent American Heart Association (AHA) emergency cardiac care guidelines suggest that there is a need to develop TOR protocols for PCPs in situations where ACLS care is not rapidly available, and call for more scientific evidence to support the implementation of such guidelines.

We derived and prospectively validated a clinical prediction rule to guide PCP termination of resuscitation in out of hospital cardiac arrest.

The TOR implementation study aims to document the usefulness of the TOR guideline, as specified by a newly developed medical directive, in decreasing the rate of transport of OHCA patients to the ED. Secondary aims of this implementation study will be to describe the rates of erroneous application of the guideline. The comfort of use of the rule among paramedics and base hospital emergency physicians will be described.

This will be a multi-centre prospective implementation study involving a combination of urban and rural regional EMS systems across Ontario. Included will be consecutive patients who suffer from non-traumatic cardiac arrest (i.e. of presumed cardiac etiology). Identical to the derivation and validation phase, patients will be excluded from the study if: their arrest is due to trauma, drowning or drug overdose; they receive any prehospital ACLS care; they possess a documented "Do Not Resuscitate" directive; or they are less than 18 years of age.

Cases that meet inclusion criteria will be enrolled consecutively. For each cardiac arrest, paramedics will respond to the call as usual and initiate resuscitation attempts. Patients suffering from cardiac arrest that (1) was not witnessed by EMS personnel; (2) had no shocks delivered by anyone; and (3) have had no return of spontaneous carotid or femoral pulse meet the criteria for TOR. In these circumstances PCPs will patch to the local BHP using the standard patching process. The BHP will then direct the paramedic to either continue resuscitation and transport, or terminate resuscitation in the field based on the TOR guideline and their clinical judgment of each individual call. In the case of failure of the paramedic to reach the BHP, the paramedic is directed to continue resuscitation and transport as per normal procedures, regardless of what the TOR guideline recommends. Data for each case will be requested from both the paramedic and the emergency physician using a uniform data collection sheet and the standardized Ontario Ambulance Call Report (ACR).

The rate of patient transport to the ED will be calculated. The obtained rate of transport will be compared to the theoretical rate obtained in the validation study, 37.4% using a one sample test, two sided, test of proportions, in order to evaluate the utility of the rule to decrease transport rates. Rates of erroneous application of the rule by both paramedics and emergency physicians will be calculated by identifying and tabulating the various reason for non-compliance. Occurrence of adverse patient outcomes, such as ROSC after TOR will be closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* No advanced cardiac life support procedures (ACLS) were available during the call
* The cardiac arrest is of presumed cardiac cause only

Exclusion Criteria:

* Age < 18
* The patient possesses a documented do-not-resuscitate (DNR) order
* The cardiac arrest is due to non cardiac causes such as trauma, drowning or drug overdose
* Patient receives any prehospital ACLS care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a multi centre prospective observational study of the implementatiaon of a Basic Life Support Termination of Resuscitation(BLS TOR)guideline.The study will accrue all out of hospital cardiac arrest cases from 9 regions across the province of Ontario(Cornwall, Hamilton,Peel, Peterborough, Grey Bruce Huron, Timmins, Sault Ste Marie, Simcoe/Muskoka, Cambridge). There are 22 participating EMS systems over the 9 regions.
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2006-01; Primary Completion 2010-12 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie J Morrison, MD, Principal Investigator — Rescu, St. Michael's Hospital Toronto; Richard P Verbeek, MD, Principal Investigator — Division of Emergency Medicine, Department of Medicine, University of Toronto and Sunnybrook Osler Center for Prehospital Care; Don Eby, MD, Principal Investigator — Grey Bruce Huron Paramedic Base Hospital Program, Grey Bruce Health Services, Owen Sound Hospital
Locations (7):
- Canada (7):
  - Royal Victoria Hospital, Barrie, Ontario
  - Cornwall Community Hospital, Cornwall, Ontario
  - Hamilton Health Sciences, Hamilton, Ontario
  - Grey Bruce Huron, Owen Sound, Ontario
  - Peterborough Regional Health Center, Peterborough, Ontario
  - Sault Area Hospital, Sault Ste. Marie, Ontario
  - Timmins and District Hospital, Timmins, Ontario

REFERENCES:
- [Background] Morrison LJ, Visentin LM, Kiss A, Theriault R, Eby D, Vermeulen M, Sherbino J, Verbeek PR; TOR Investigators. Validation of a rule for termination of resuscitation in out-of-hospital cardiac arrest. N Engl J Med. 2006 Aug 3;355(5):478-87. doi: 10.1056/NEJMoa052620. PMID 16885551
- [Background] Verbeek PR, Vermeulen MJ, Ali FH, Messenger DW, Summers J, Morrison LJ. Derivation of a termination-of-resuscitation guideline for emergency medical technicians using automated external defibrillators. Acad Emerg Med. 2002 Jul;9(7):671-8. doi: 10.1111/j.1553-2712.2002.tb02144.x. PMID 12093706
- [Background] Morrison LJ, Cheung MC, Redelmeier DA. Evaluating paramedic comfort with field pronouncement: development and validation of an outcome measure. Acad Emerg Med. 2003 Jun;10(6):633-7. doi: 10.1111/j.1553-2712.2003.tb00047.x. PMID 12782524
- [Background] Morrison LJ, Visentin LM, Vermeulen M, Kiss A, Theriault R, Eby D, Sherbino J, Verbeek R; TOR investigators. Inter-rater reliability and comfort in the application of a basic life support termination of resuscitation clinical prediction rule for out of hospital cardiac arrest. Resuscitation. 2007 Jul;74(1):150-7. doi: 10.1016/j.resuscitation.2006.10.030. Epub 2007 Feb 14. PMID 17303311
- [Background] Morrison LJ, Verbeek PR, Vermeulen MJ, Kiss A, Allan KS, Nesbitt L, Stiell I. Derivation and evaluation of a termination of resuscitation clinical prediction rule for advanced life support providers. Resuscitation. 2007 Aug;74(2):266-75. doi: 10.1016/j.resuscitation.2007.01.009. Epub 2007 Mar 23. PMID 17383072